CLINICAL TRIAL: NCT04160338
Title: A Specular Microscopic Study of Corneal Endothelium After Accelerated Corneal Collagen Cross Linking
Brief Title: Assessment of Corneal Endothelium After Collagen Cross Linking
Acronym: CXL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Naglaa Mostafa Abdelhafez Abdelmohsen, resident doctor, Assiut University
Other Study IDs: corneal collagen cross linking
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Accelerated Corneal Collagen Cross Linking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: specular microscopy — An informed written consent will be obtained from all patients that will be included in this study. Patients in this study will undergo specular microscopic examination of corneal endothelium before CXL procedure.
  Patients will be assigned to undergo accelerated (epithelium-off ,transepithelial ) CXL .
  Follow up specular microscopy will be done 3 months and 6 months after corneal collagen cross linking procedure .

SUMMARY:
The aim of this study is to assess the effect of accelerated corneal collagen cross linking on corneal endothelium using the specular microscopy

DETAILED DESCRIPTION:
Keratoconus (KC) is a progressive, non-inflammatory corneal degenerative disease. It is a pathology characterized by a progressive thinning and protrusion of the cornea that ends in a cone-shaped cornea. This results in progressive myopia and irregular astigmatism with associated progressive loss of vision and thus reduced quality of life.Collagen cross-linking (CXL) is a relatively new conservative approach for progressive corneal ectasia. The main indication for CXL is to slow the progression of corneal ectatic diseases, such as keratoconus, pellucid marginal degeneration (PMD), keratoglobus and iatrogenic ectasia.The basic principle of this method is the chemical interaction of ultraviolet A radiation (315-400nm ) and riboflavin to induce covalent bond formation between collagen fibers of the cornea. In this way, the stiffness and rigidity of the cornea are provided.Corneal collagen cross-linking (CXL) was first introduced by Wollensak with an ultraviolet-A (UVA) protocol of 3 medium wave mW/cm2 intensity at 370 nm over an exposure time of 30 minutes (now termed the "Dresden protocol"). Researchers have proposed accelerated CXL (ACXL) protocols, to improve convenience and comfort for patients. These ACXL protocols have the aim of decreasing UVA exposure time by increasing UVA fluency to achieve the same overall total UVA dosage.Despite corneal CXL is a safe and effective procedure with few known side effects .Persistent corneal edema and possible endothelial cell damage have been reported in a few cases after CXL. Based on the extent of endothelial damage, patients may require penetrating keratoplasty.

ELIGIBILITY:
Inclusion Criteria:

1. patients with mild to moderate corneal ectasia who are candidates for CXL.

Exclusion Criteria:

1. patients with advanced corneal ectasia with maximum keratometry readings <56 diopters.
2. corneal pachymetry >380um.
3. corneal scarring.
4. previous corneal surgeries (e.g intrastromal corneal ring segments)

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients who underwent accelerated corneal collagen cross linking
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
endothelial cell count by specular microscopy. | from preoperatively to 6 months postoperatively
  specular microscopy will be used to assess corneal endothelial cell count after accelerated corneal collagen cross linking

SECONDARY OUTCOMES:
endothelial cell morphology by specular microscopy. | from preoperatively to 6 months postoperatively
  specular microscopy will be used to assess corneal endothelial cell morphology after accelerated corneal collagen cross linking

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed T Abdelmonem, Professor, Study Director — Assiut Uneversity; Hazem A Hazem, lecturer, Study Director — Assiut Uneversity; Mahmoud A Abdelsalam, lecturer, Study Director — Assiut Uneversity

REFERENCES:
- [Background] Raiskup-Wolf F, Hoyer A, Spoerl E, Pillunat LE. Collagen crosslinking with riboflavin and ultraviolet-A light in keratoconus: long-term results. J Cataract Refract Surg. 2008 May;34(5):796-801. doi: 10.1016/j.jcrs.2007.12.039. PMID 18471635
- [Background] Subasinghe SK, Ogbuehi KC, Dias GJ. Current perspectives on corneal collagen crosslinking (CXL). Graefes Arch Clin Exp Ophthalmol. 2018 Aug;256(8):1363-1384. doi: 10.1007/s00417-018-3966-0. Epub 2018 Apr 6. PMID 29623463
- [Background] Mencucci R, Marini M, Paladini I, Sarchielli E, Sgambati E, Menchini U, Vannelli GB. Effects of riboflavin/UVA corneal cross-linking on keratocytes and collagen fibres in human cornea. Clin Exp Ophthalmol. 2010 Jan;38(1):49-56. doi: 10.1111/j.1442-9071.2010.02207.x. PMID 20447101
- [Background] Wen D, Li Q, Song B, Tu R, Wang Q, O'Brart DPS, McAlinden C, Huang J. Comparison of Standard Versus Accelerated Corneal Collagen Cross-Linking for Keratoconus: A Meta-Analysis. Invest Ophthalmol Vis Sci. 2018 Aug 1;59(10):3920-3931. doi: 10.1167/iovs.18-24656. PMID 30073363
- [Background] Kirgiz A, Eliacik M, Yildirim Y. Different accelerated corneal collagen cross-linking treatment modalities in progressive keratoconus. Eye Vis (Lond). 2019 Jun 3;6:16. doi: 10.1186/s40662-019-0141-6. eCollection 2019. PMID 31172016
- [Background] Zhang X, Zhao J, Li M, Tian M, Shen Y, Zhou X. Conventional and transepithelial corneal cross-linking for patients with keratoconus. PLoS One. 2018 Apr 5;13(4):e0195105. doi: 10.1371/journal.pone.0195105. eCollection 2018. PMID 29621306
- [Background] Vazirani J, Bagga B, Taneja M. Persistent corneal edema after collagen cross-linking for keratoconus. Am J Ophthalmol. 2013 Apr;155(4):775. doi: 10.1016/j.ajo.2013.01.003. No abstract available. PMID 23521904
- [Background] Sedaghat M, Bagheri M, Ghavami S, Bamdad S. Changes in corneal topography and biomechanical properties after collagen cross linking for keratoconus: 1-year results. Middle East Afr J Ophthalmol. 2015 Apr-Jun;22(2):212-9. doi: 10.4103/0974-9233.151877. PMID 25949080
- [Derived] Abdel-Radi M, Abdelmohsen N, Abdelmotaal H, Abd El-Moneim MT. The effect of accelerated pulsed high-fluence corneal cross-linking on corneal endothelium; a prospective specular microscopy study. BMC Ophthalmol. 2023 Apr 18;23(1):163. doi: 10.1186/s12886-023-02912-6. PMID 37072730